CLINICAL TRIAL: NCT00056797
Title: A Randomized Controlled Study Testing the Efficacy of Immunotherapies to Control Plasma HIV RNA Concentrations Upon Interruption of Highly Active Antiretroviral Therapy (HAART).
Brief Title: Therapeutic HIV Vaccine and Interleukin-2 to Increase the Immune System's Response to HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AI051181-01A1 (NIH); 0900-397; 1R01AI051181-01A1 (NIH)
Record Dates: First submitted 2003-03-24; First posted 2003-03-25 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infections
Keywords: HIV Therapeutic vaccine; IL-2; Structured Treatment Interruption; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2

INTERVENTIONS:
Biological: ALVAC HIV vaccine (vCP1452)
Drug: Interleukin-2

SUMMARY:
This study will evaluate whether the HIV vaccine ALVAC vCP1452 given in combination with interleukin-2 (IL-2), also known as aldesleukin, can increase immune system function in people with HIV infection.

DETAILED DESCRIPTION:
While the advent of highly active antiretroviral therapy (HAART) has contributed to the increasing control of HIV infection and viral replication, ultimate control of HIV infection will require the development of effective HIV-specific immunity in HIV infected individuals.

This trial will evaluate the use of the ALVAC vCP1452 vaccine in combination with IL-2 to increase HIV-specific immune responses in HIV infected patients. ALVAC vCP1452 vaccine is a recombinant canarypox HIV vaccine that is administered as a monthly intramuscular injection. The IL-2 is self administered as a daily subcutaneous injection at a low, non-toxic dose (2 million units).

Participants in this study are randomized to receive either ALVAC and IL-2 or placebo for the first 3 months of the study. During this time, participants will continue on their current antiretroviral medications and have monthly study visits. Study visits will include a brief medical interview and physical exam, administration of the vaccine, and blood tests. At the end of 3 months, participants will discontinue both their study medications (IL-2 and ALVAC or placebo) and their antiretroviral medications. This Diagnostic Treatment Interruption (DTI) will continue for a minimum of 3 months. During the DTI, participants will have weekly study visits in which viral and lymphocyte dynamics are monitored.

ELIGIBILITY:
Inclusion Criteria

* HIV infected
* Stable HAART, defined as two or more antiretroviral drugs in combination. Changes in drugs are allowed if for any reason other than virologic failure.
* CD4 cell count > 200 cells/ml for the 12 months prior to enrollment
* CD4 cell count >= 400 cells/ml on two successive occasions at least 14 days apart within 30 days of study entry
* HIV RNA < 2 million copies/ml, with suppression on HAART to < 50 copies/ml on two successive occasions at least 14 days apart within 30 days of entry
* Acceptable methods of contraception

Exclusion Criteria

* Current AIDS-defining illness
* Virologic failure (HIV RNA > 10,000 copies/ml) while receiving current HAART regimen
* Immunomodulating agents, including interleukins; antibodies reactive with lymphocytes, monocytes, or antigen presenting cells; and polyribonucleotides
* IL-2 therapy within 4 weeks of study entry
* Uncontrolled active cardiac, renal, pulmonary, hepatic, or CNS disease
* History of active malignancy requiring chemotherapy
* History of thyroid disease or autoimmune disorders, including asthma, inflammatory bowel disease, rheumatoid arthritis, and psoriasis
* Active infection with hepatitis B virus or hepatitis C virus
* Severe retinopathy due to diabetes, hypertension, CMV, or macular degeneration
* Serious infection or other serious medical illness that is potentially life threatening and requires systemic therapy and/or hospitalization within 14 days of study entry
* Substance abuse that will compromise the participant's ability to adhere to the study requirements
* Current alcohol use of more than 1 drink/day any time during 6 months prior to study entry. One drink is defined as 12 ounces of beer, 5 ounces of wine, or 1.25 ounces of hard liquor.
* History of allergy to eggs, IL-2, or other components of the vaccine or IL-2 formulation
* Pregnant or breast-feeding
* Professionals working in close contact with canaries (e.g., breeding farms, bird shops)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92
Dates: Start 2002-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Mean log10 viral load for each experimental group from the average of 5 values obtained during Weeks 21 to 25, corresponding to 8 to 12 weeks following the interruption of HAART

SECONDARY OUTCOMES:
Proportion of subjects who relapse during the first 12 weeks following cessation of HAART
length of time to the termination of Step II
changes in frequency, activation state, and HIV-specific functional capacity of T cells and NK cells in blood, as monitored by the expression of intracellular cytokines during the first 12 weeks after cessation of HAART

CONTACTS AND LOCATIONS:
Overall Officials: Kendall A. Smith, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NY Presbyterian Weill Cornell Medical Center, New York, New York, United States